CLINICAL TRIAL: NCT07390942
Title: Tongue and Occlusal Pressure Performance and Dietary Habits in Maxillectomy Patients With Obturator Prostheses
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202507230RINC
Record Dates: First submitted 2025-11-17; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Maxillary Obturators; Maxillary Defect Reconstruction; Dietary Behavior
Keywords: Obturator; Dental Prescale II; EAT-10; Tongue pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maxillectomy patients with obturator prosthesis

SUMMARY:
This study investigates mouth cancer patients who use a special plate called an obturator to help them swallow. Tongue strength and biting force will be measured and compared to daily dietary intake. Results will provide a better understanding of how to improve eating ability and overall quality of life.

DETAILED DESCRIPTION:
For oral cancer patients who have undergone maxillectomy, the use of an obturator can help restore partial swallowing function, thereby improving quality of life. Measuring tongue pressure provides insight into the extent of a patient's swallowing function, while occlusal pressure measurement assesses occlusal force, offering guidance for dietary modifications. This study will utilize a tongue pressure measurement device and occlusal pressure Prescale film to quantify tongue elevation pressure and occlusal force in post-maxillectomy oral cancer patients who wear obturators. This will be complemented by questionnaires to understand the participants' daily dietary habits and content. The aim is to establish the distribution of tongue and bite pressures within this patient population and to preliminarily determine the correlation between these pressures and daily diet

ELIGIBILITY:
Inclusion Criteria:

* Primary treatment must include maxillectomy, with or without adjuvant chemotherapy or radiotherapy.
* Age range: 18 to 85 years old (all genders).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Ability to provide written informed consent.

Exclusion Criteria:

* Inability to understand the investigator's instructions (or indications).
* Inability to hold the tongue pressure probe and occlusal pressure Prescale film in the proper position.
* Inability to apply pressure to the tongue pressure probe and occlusal pressure Prescale film.
* Dysphagia (difficulty swallowing) resulting from prior head and neck cancer treatment.
* Severe dysphagia caused by a central nervous system disorder.
* Presence of temporomandibular joint (TMJ) pain.
* The investigator determines the patient is unsuitable for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical trial will be conducted at the Outpatient Department of Dentistry at National Taiwan University Hospital.
  The study subjects will be oral cancer patients who have undergone maxillectomy and wear an obturator. They will be recruited from patients routinely followed up and treated by the principal investigator, or similar patients referred by colleagues within the same department.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tongue Pressure | Baseline
  Tongue pressure is measured using the Iowa Oral Performance Instrument (IOPI). The pressure balloon is positioned on either the anterior tongue (behind the anterior alveolar ridge) or the posterior tongue (at the junction of the hard and soft palate). The subject is instructed to press the pressure balloon firmly with their tongue for a duration of 2 seconds. The procedure is repeated three times after a 30-60 second rest period. The maximum pressure value obtained will be recorded.
  Unit of Measure: kilopascals (kPa)
Maximum Occlusal Force | Baseline
  Occlusal force is measured using the Prescale II film. An appropriate size of the film is placed into the mouth, ensuring occlusal surfaces are within the area. The subject is asked to bite down firmly for 3 seconds. The film is then scanned using a dedicated scanner, and specialized software performs image processing to quantify the occlusal force.
  Unit of Measure: Newtons (N)

SECONDARY OUTCOMES:
Eating Assessment Tool-10 (EAT-10) Score | Baseline
  The traditional Chinese version of the EAT-10 is used to assess swallowing dysphagia symptom severity. It consist of 10 questions, each scored from 0 (no problem) to 4 (severe problem). The total score ranges from 0 to 40, with higher scores indicating higher self-perception of swallowing impairment.
  Unit of Measure: Score on a scale
Daily Meal Frequency | Baseline
  Participants report the number of meals consumed on the previous day using a 5-category scale (1, 2, 3, 4, or 5 or more meals).
  Unit of Measure: Number of meals per day
Dietary Food Texture Consumption | Baseline
  Participants identify the texture levels of the foods they currently consume based on the IDDSI (International Dysphagia Diet Standardisation Initiative) framework, ranging from Level 0 to Level 7. Multiple levels may be selected to reflect their dietary range.
  Unit of Measure: Percentage of participants reporting each texture level
Frequency of Dining Out | Baseline
  Participants report their frequency of eating out (including food delivery) on a 5-point ordinal scale (Always, Mostly, Frequently, Occasionally, Never).
  Unit of Measure: Percentage of participants per frequency category
Self-Reported Pronunciation Difficulty | Baseline
  Participants rate their ease of pronunciation using a 4-point ordinal scale: Normal (1), Slightly inconvenient (2), A bit difficult (3), and Very difficult (4).
  Unit of Measure: Score on a scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dentistry of National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Raw Dataset Baseline Characteristics Outcome Measures
Supporting Information: Study Protocol, ICF
Time Frame: 9 months after the end of strudy and last until 24 months

REFERENCES:
- [Result] Wang TM, Chang YH, Yang TC, Lin LD. Effect of scan delay on measurements of an occlusal pressure sensitive film: An in-vitro study. J Dent Sci. 2022 Jan;17(1):30-34. doi: 10.1016/j.jds.2021.08.005. Epub 2021 Aug 28. PMID 35028017
- [Result] Clark HM, Solomon NP. Age and sex differences in orofacial strength. Dysphagia. 2012 Mar;27(1):2-9. doi: 10.1007/s00455-011-9328-2. Epub 2011 Feb 25. PMID 21350818
- [Result] Vanderwegen J, Guns C, Van Nuffelen G, Elen R, De Bodt M. The influence of age, sex, bulb position, visual feedback, and the order of testing on maximum anterior and posterior tongue strength and endurance in healthy belgian adults. Dysphagia. 2013 Jun;28(2):159-66. doi: 10.1007/s00455-012-9425-x. Epub 2012 Sep 16. PMID 22983359
- [Result] Zhang PP, Yuan Y, Lu DZ, et al. Diagnostic Accuracy of the Eating Assessment Tool-10 (EAT-10) in Screening Dysphagia: A Systematic Review and Meta-Analysis. Dysphagia. 2023;38(1):145-158.
- [Result] Matsuyama M, Tsukiyama Y, Tomioka M, Koyano K. Clinical assessment of chewing function of obturator prosthesis wearers by objective measurement of masticatory performance and maximum occlusal force. Int J Prosthodont. 2006 May-Jun;19(3):253-7. PMID 16752621
- [Result] Shiga H, Komino M, Yokoyama M, et al. Relationship between age and occlusal force in adults with natural dentition. Odontology. 2023;111(2):487-492.
- [Result] Miura H, Watanabe S, Isogai E, Miura K. Comparison of maximum bite force and dentate status between healthy and frail elderly persons. J Oral Rehabil. 2001;28(6):592-595.
- [Result] Van den Steen L, Vanderveken O, Vanderwegen J, et al. Member of the Belgian Cancer Plan 29_033_Dysphagia Group. Feasibility of tongue strength measurements during (chemo) radiotherapy in head and neck cancer patients. Support Care Canc 2017;25:3417-23.
- [Result] Lazarus CL, Logemann JA, Pauloski BR, et al. Swallowing and tongue function following treatment for oral and oropharygeal cancer. J Speech Lang Hear Res 2000;43:1011-23.
- [Result] Tanaka A, Uemura H, Kimura T, et al. Evaluation of usefulness of tongue pressure measurement device for dysphagia associated with treatment of patients with head and neck cancer (ELEVATE). Medicine (Baltimore). 2023;102(26):e33954.
- [Result] Adams V, Mathisen B, Baines S, Lazarus C, Callister R. Reliability of measurements of tongue and hand strength and endurance using the Iowa Oral Performance Instrument with healthy adults. Dysphagia. 2014 Feb;29(1):83-95. doi: 10.1007/s00455-013-9486-5. Epub 2013 Sep 18. PMID 24045852
- [Result] Brown JS, Shaw RJ. Reconstruction of the maxilla and midface: introducing a new classification. Lancet Oncol. 2010 Oct;11(10):1001-8. doi: 10.1016/S1470-2045(10)70113-3. PMID 20932492